CLINICAL TRIAL: NCT00781768
Title: Prevention of Nausea and Vomitting Associated With Stem Cell Transplant: Results of a Prospective, Randomized Trial of Aprepitant Used With Highly Emetogenic Preparative Regimens
Brief Title: Odansetron and Dexamethasone Alone vs. Odansetron, Dexamethason and Apreptant to Prevent Nausea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Patrick Stiff, Professor and Director of the Cardinal Bernardin Cancer Center, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 106578
Record Dates: First submitted 2008-10-27; First posted 2008-10-29 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Nausea; Vomiting
Keywords: Bone Marrow Transplant; Nausea; Vomiting; NK-1 antagonist
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron; Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard PO (Zofran + Dexamethasone) (Placebo Comparator): Dexamethasone 10 mg (dose blinded) in 50 ml D5W IVPB over 15 minutes daily + ondansetron (Zofran) 8mg PO q 8 hours - repeated qd of the preparative regimen and for 1 day after completion.
  Interventions: Drug: Standard PO (Zofran + Dexamethason)
- Aprepitant (MK-869) + Standard PO (Active Comparator): Dexamethasone 7.5 mg (dose blinded) in 50 ml D5W IVPB over 15 min daily + ondansetron 8mg PO q 8 hours - repeated QD of the preparative regimen and for 1 day after completion. Aprepitant 125mg PO [blinded] will be given a minimum of 30 minutes prior to the preparative regimen on day 1. MK-Aprepitant 80mg PO [blinded] will be given will be given approximately 24 hours later starting on day 2 then each day of the preparative regimen plus 3 days after. Antiemetic therapy will start a minimum of 30 minutes prior to and continued for 24 hours after completion of the preparative regimen.
  Interventions: Drug: Aprepitant (MK-869) + Standard PO

INTERVENTIONS:
Drug: Standard PO (Zofran + Dexamethason) — Dexamethasone 10 mg (dose blinded) in 50 ml D5W IVPB over 15 minutes daily + ondansetron 8mg PO q 8 hours - repeated qd of the preparative regimen and for 1 day after completion. A placebo capsule will be given daily on each day of the preparative regimen plus 3 days after. Antiemetic therapy will start a minimum of 30 minutes prior to and continued for 24 hours after completion of the preparative regimen.
  Other Names: Ondansetron (Zofran)
  Arms: Standard PO (Zofran + Dexamethasone)
Drug: Aprepitant (MK-869) + Standard PO — Dexamethasone 7.5 mg (dose blinded) in 50 ml D5W IVPB over 15 min daily + ondansetron 8mg PO q 8 hours - repeated QD of the preparative regimen and for 1 day after completion. Aprepitant 125mg PO [blinded] will be given a minimum of 30 minutes prior to the preparative regimen on day 1. MK-Aprepitant 80mg PO [blinded] will be given will be given approximately 24 hours later starting on day 2 then each day of the preparative regimen plus 3 days after. Antiemetic therapy will start a minimum of 30 minutes prior to and continued for 24 hours after completion of the preparative regimen.
  Other Names: Ondansetron + Dexamethason (Standard PO)
  Arms: Aprepitant (MK-869) + Standard PO

SUMMARY:
The purpose of this study is to compare two different treatment protocols for treating nausea and vomiting in patients who have undergone bone marrow transplant. Patients will be assigned to one of two treatment groups.

The first group will recieve ondansetron (Zofran) tablets combined with a medicine called dexamethasone given IV. Both of these drugs are commercially available.

Patients in the second treatment consists of the first two drugs, plus a newly approved drug known as aprepitant (MK-869, Emend). This combination will be the treatment being tested. The combination is approved by the FDA for chemotherapy regimens known to cause a lot of nausea and vomiting. It significantly decreases the delayed (more than 24 hours after therapy) nausea and vomiting seen with these regimens.

DETAILED DESCRIPTION:
This will be a single center, comparative, randomized, double-blind, phase III trial designed to evaluate the efficacy of the NK-1 antagonist, aprepitant (MK-869), in combination with ondansetron and dexamethasone in the prevention of acute and delayed nausea and vomiting compared to ondansetron and dexamethasone in patients receiving highly emetogenic preparative regimens prior to autologous or allogeneic (related and unrelated) stem cell transplantation.

Patients will be randomized to one of two treatments: dexamethasone 10 mg IV once daily and ondansetron 8 mg orally every 8 hours on each day of the preparative regimen plus one additional day vs. 7.5 mg IV once daily and ondansetron 8 mg orally every 8 hours on each day of the preparative regimen plus one additional day combined with aprepitant, 125 mg orally on the first day of their preparative regimen followed by 80 mg daily on each remaining day of the preparative regimen plus three additional days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer, admitted for myelosupppresive stem cell transplantation. Included preparative regimens include: TBI/VP16/CY, TBI/CY, BU/CY (PO & IV), and BCV
* Age 18 or older
* Alcohol intake <100 gm/d for the last year (< approximately 5 drinks per day)
* Renal function: estimated or measured CrCl 50 ml/min
* Liver function: T.Bili <1.5, AST < 2x ULN, unless due to disease
* Able to swallow tablets and capsules

Exclusion Criteria:

* Age < 18
* High alcohol intake [> 100 gm/d in the last year]
* Allergy or intolerance to: ondansetron or dexamethasone
* Renal dysfunction [measured or estimated CrCl < 50 ml/min]
* Liver dysfunction [T.Bili > 1.5, AST > 2x ULN, unless due to disease]
* Inability to swallow tablets or capsules
* Concurrent condition requiring systemic steroid use
* Nonmyeloablative SCT, patients receiving the conditioning regimens not included [see inclusion criteria]
* History of anticipatory nausea and vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2003-08; Primary Completion 2008-10 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stiff, MD, Principal Investigator — Loyola University Cardinal Bernadin Cancer Center

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard PO Ondanestron + Dexamethason: Dexamethasone 10 mg (dose blinded) in 50 ml D5W IVPB over 15 minutes daily + ondansetron 8mg PO q 8 hours - repeated qd of the preparative regimen and for 1 day after completion. A placebo capsule will be given daily on each day of the preparative regimen plus 3 days after. Antiemetic therapy will start a minimum of 30 minutes prior to and continued for 24 hours after completion of the preparative regimen.
- Aprepitant (MK-869) + Standard PO Ondanestron + Dexamethason: Dexamethasone 7.5 mg (dose blinded) in 50 ml D5W IVPB over 15 min daily + ondansetron 8mg PO q 8 hours - repeated QD of the preparative regimen and for 1 day after completion. Aprepitant 125mg PO [blinded] will be given a minimum of 30 minutes prior to the preparative regimen on day 1. MK-Aprepitant 80mg PO [blinded] will be given will be given approximately 24 hours later starting on day 2 then each day of the preparative regimen plus 3 days after. Antiemetic therapy will start a minimum of 30 minutes prior to and continued for 24 hours after completion of the preparative regimen.
Period: Overall Study
Arm/Group | Standard PO Ondanestron + Dexamethason | Aprepitant (MK-869) + Standard PO Ondanestron + Dexamethason
Started | 89 | 92
Completed | 89 | 90
Not Completed | 0 | 2
Not completed — Not transplanted. | 0 | 2

BASELINE CHARACTERISTICS:
Population: Autologous and allogeneic hematopoietic stem cell transplant patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard PO Ondanestron + Dexamethason | Aprepitant (MK-869) + Standard PO Ondanestron + Dexamethason | Total
Number analyzed (Participants) | 89 | 90 | 179
Age, Continuous [Median (Full Range); unit: years] | 51 [19 to 79] | 50 [20 to 75] | 50 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 57 | 57 | 114
Diagnosis [Count of Participants; unit: Participants]
  Non-Hodgkin lymphoma | 28 | 29 | 57
  Acute Myelogenous Leukemia | 22 | 24 | 46
  Multiple Myeloma | 21 | 13 | 34
  Acut Lymphoblastic Lymphoma | 3 | 10 | 13
  Hodgkin's lymphoma | 7 | 5 | 12
  Chronic Myelogenous Leukemia | 4 | 2 | 6
  Other | 4 | 7 | 11
Setting [Count of Participants; unit: Participants]
  Inpatient | 69 | 74 | 143
  Outpatient | 20 | 16 | 36
Graft Type [Count of Participants; unit: Participants]
  Autologous-peripheral blood stem cell transplant | 48 | 41 | 89
  Related Allo-PBPCT | 19 | 22 | 41
  Related autologous bone marrow transplant | 1 | 1 | 2
  Matched unrelated donor PBPCT | 8 | 12 | 20
  Matched unrelated donor BMT | 6 | 8 | 14
  Cord as in umbilical cord | 7 | 6 | 13
Preparative Regimen [Count of Participants; unit: Participants]
  Total body irradiation/Cyclophosphamide | 33 | 46 | 79
  I.V. Busulfan/Cy | 7 | 7 | 14
  Prescribed orally Bu/Cy | 21 | 13 | 34
  TBI/Etoposide/Cy | 17 | 19 | 36
  BCV | 11 | 5 | 16
History of prior nausea or vomiting with chemotherapy [Count of Participants; unit: Participants]
  Yes | 55 | 59 | 114
  No | 30 | 25 | 55
  Unknown | 4 | 6 | 10
History of prior nausea or vomiting with radiation therapy [Count of Participants; unit: Participants]
  Yes | 42 | 41 | 83
  No | 43 | 42 | 85
  Unknown | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rates Among Standard of Care and Combination Therapy Groups.
Description: Comparison of complete response (CR) rates between patients receiving ondansetron and dexamethasone and those receiving ondansetron and dexamethasone plus NK-1 antagonist, aprepitant. CR is defined as no emesis and with normal oral intake. Disease response not applicable.
Time Frame: 14 days
Population: 179 patients receiving autologous and allogeneic hematopoietic stem cell transplants.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard PO Ondanestron + Dexamethason | Aprepitant (MK-869) + Standard PO Ondanestron + Dexamethason
Number analyzed (Participants) | 89 | 90
Participants
  Complete Responder | 58 | 73
  Not Complete Responder | 31 | 17
Statistical Analysis 1: Comparison: Standard PO Ondanestron + Dexamethason vs Aprepitant (MK-869) + Standard PO Ondanestron + Dexamethason; The null hypothesis is that there will be a higher proportion of complete responders among those subjects receiving the combination therapy; Test type: Superiority; p < .001, Chi-squared; Odds Ratio (OR) = 2.30

ADVERSE EVENTS:
Time Frame: Adverse events data were collected through study completion, or 7 years.
Arm/Group | Standard PO Ondanestron + Dexamethason | Aprepitant (MK-869) + Standard PO Ondanestron + Dexamethason
All-Cause Mortality (participants affected / at risk) | 2/89 | 5/90
Serious Adverse Events (participants affected / at risk) | 2/89 | 5/90
Other Adverse Events (participants affected / at risk) | 52/89 | 59/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard PO Ondanestron + Dexamethason (N=89) | Aprepitant (MK-869) + Standard PO Ondanestron + Dexamethason (N=90)
Sepsis (Infections and infestations) | 0 (0) | 4 (4)
Veno-occlusive disease of the liver (Infections and infestations) | 0 (0) | 1 (1)
Viral Pneumonia/Encephalitis and fungal Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard PO Ondanestron + Dexamethason (N=89) | Aprepitant (MK-869) + Standard PO Ondanestron + Dexamethason (N=90)
Diarrhea (Gastrointestinal disorders) | 52 (52) | 59 (59)
Headache (General disorders) | 46 (46) | 44 (44)
Fatigue (General disorders) | 34 (34) | 37 (37)
Constipation (Gastrointestinal disorders) | 21 (21) | 28 (28)
Fever (General disorders) | 19 (19) | 22 (22)
Hiccups (General disorders) | 20 (20) | 21 (21)
Heartburn (Gastrointestinal disorders) | 6 (6) | 12 (12)
Lightheartedness/dizziness (General disorders) | 5 (5) | 7 (7)

LIMITATIONS AND CAVEATS:
There are no limitations or caveats to disclose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes